CLINICAL TRIAL: NCT03830112
Title: Effects of a Pilates-based Mat Exercise Program Compared to a Pilates-based Mat Exercise With Resistance Band on the Isometric Strength of Core Muscles, Lean Mass, and Body Fat in Men 18 to 25 Years
Brief Title: Effect of Two Pilates-based Mat Exercise Programs on the Isometric Strength of Core Muscles in Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Victor Hugo Arboleda Serna, Associate Professor, Universidad de Antioquia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mat Pilates
Record Dates: First submitted 2019-02-01; First posted 2019-02-05 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercise with Theraband (Experimental): 24 exercise sessions, 3x weekly (on alternate days).
  11 Pilates-based exercises with Theraband® (blue color) from week one to four. (hundred,roll up, one leg circle,rolling like a ball,single leg stretch, double leg stretch,single straight leg stretch, double straight leg lower lift, criss-cross, spine stretch, corkscrew).
  12 Pilates-based exercises with Theraband® (blue color) from week five to eight.
  (saw, rest position, shoulder bridge, side, kick, front ad back, up and down, teaser, swimming, leg pull front, mermaid, seal, push up).
  Every participant will perform three isometric repetitions of 30 seconds per exercise, with 10 seconds recovery between repetitions and 30 seconds rest between each exercise.
  Interventions: Behavioral: Pilates exercise with Theraband
- Pilates exercise (Active Comparator): 24 exercise sessions, 3x weekly (on alternate days).
  11 Pilates-based mat exercises from week one to four. (hundred,roll up, one leg circle,rolling like a ball,single leg stretch, double leg stretch,single straight leg stretch, double straight leg lower lift, criss-cross, spine stretch, corkscrew).
  12 Pilates-based mat exercises from week five to eight. (saw, rest position, shoulder bridge, side, kick, front ad back, up and down, teaser, swimming, leg pull front, mermaid, seal, push up).
  Every participant will perform three isometric repetitions of 30 seconds per exercise, with 10 seconds recovery between repetitions and 30 seconds rest between each exercise.
  Interventions: Behavioral: Pilates exercise

INTERVENTIONS:
Behavioral: Pilates exercise with Theraband — The experimental group will perform all the exercises with Theraband® in the same manner than active comparator group.
  Arms: Pilates exercise with Theraband
Behavioral: Pilates exercise — The active comparator group will perform all the exercises without Theraband®
  Arms: Pilates exercise

SUMMARY:
Based on the current evidence, it is known that Pilates is an exercise technique that has been used mainly by women in sport, fitness and rehabilitation. Most research has been developed with women. The participation of men in the research studies is reduced and methodology rigor is low, therefore, there is insufficient evidence on the effects of this type of training in men, in addition, there are no studies that have proven the effects of a Pilates-based mat exercise with resistance band on strength of core muscles.

The main objective of this research is to identify the effects of a Pilates-based mat exercise program versus a Pilates-based exercise mat program with resistance band on the isometric strength of the core muscles in men 18 to 25 years.

DETAILED DESCRIPTION:
Fifty-eight men will be randomly assigned to one of two Pilates exercise programs. Pilates-based mat exercise and Pilates-based mat exercise with Theraband® (blue color). Interventions will be performed three times a week for eight-weeks on alternate days. Half will perform Pilates-based mat exercise and the remaining 29 will perform Pilates-based mat exercise with Theraband®. Both groups complete eleven exercises from week one to four and twelve exercises from week five to eight.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers.
* Perform ≤150 minutes of aerobic exercise per week.

Exclusion Criteria:

* Perform any Pilates exercise previously.
* Smoker.
* History of asthma.
* History of diabetes.
* History of hypertension.
* History of cardiovascular disease.
* History of coronary heart disease.
* Arrhythmias.
* Under medical treatment with anticoagulants, beta-blockers, calcium antagonists, bronchodilators, and/or steroids.
* Psychological, neuromotor and/or osteo-muscular conditions that may affect participation in an exercise program.
* People with metal prosthesis.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Change in isometric strength of the core muscles | Baseline and after 8 weeks
  Isometric strength of the core muscles will be obtained using TorsoCheck (Ergo-Fit®, Germany).

SECONDARY OUTCOMES:
Change in lean mass | Baseline and after 8 weeks
  Lean mass will be obtained using Bioelectrical impedance (SECA mBCA515, Gmbh&Co.,Hamburg,Germany)
Change in body fat | Baseline and after 8 weeks
  Body fat will be obtained using Bioelectrical impedance (SECA mBCA515,Gmbh&Co.,Hamburg,Germany).

CONTACTS AND LOCATIONS:
Overall Officials: Víctor H Arboleda Serna, PhD, Principal Investigator — Universidad de Antioquia
Locations (1):
- Centro de Formación en Actividad Física y Cultura, Bogotá, Cundinamarca, Colombia